CLINICAL TRIAL: NCT06399237
Title: Biomechanical Effects of Three Types of Foot Orthoses in Individuals With Posterior Tibialis Tendon Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Philippe Corbeil, Full Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MP-20-2018-4003
Record Dates: First submitted 2021-04-08; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Posterior Tibial Tendon Dysfunction
Keywords: Posterior tibialis tendon dysfunction, Foot orthoses,
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No orthoses (No Intervention): Walk at a self-selected pace without orthoses.
- Prefabricated foot orthoses (PFO) (Active Comparator): Walk at a self-selected pace with prefabricated foot orthoses (PFO).
  Interventions: Device: Foot Orthoses
- Custom-fitted orthoses (CFO) (Active Comparator): Walk at a self-selected pace with custom-fitted orthoses (CFO)
  Interventions: Device: Foot Orthoses
- Custom-fitted orthoses with a 5deg varus (CFVO) (Active Comparator): Walk at a self-selected pace with custom-fitted orthoses with a 5deg varus (CFVO)
  Interventions: Device: Foot Orthoses

INTERVENTIONS:
Device: Foot Orthoses — Three types of foot orthoses (FO), Prefabricated FO, Custom FO, Custom with a 5° varus FO
  Other Names: Foot Orthosis
  Arms: Custom-fitted orthoses (CFO); Custom-fitted orthoses with a 5deg varus (CFVO); Prefabricated foot orthoses (PFO)

SUMMARY:
Background :

Posterior tibialis tendon dysfunction (PTTD) is characterized by a loss of function of the muscle caused by the degeneration of the tendon leading to a flattening of the arch. FOs can be used as a treatment option, but their biomechanical effects are not yet fully understood. The aim of this study was to investigate the effects of three different types of foot orthoses (FOs) on gait biomechanics in individuals suffering from PTTD.

Methods :

Fourteen individuals were recruited with painful stage 1 or 2 PTTD based on the Johnson and Strom's classification. Quantitative gait analysis of the affected limb was performed in four conditions: shoed condition (Shoe), prefabricated FOs condition (PFO), neutral custom FOs condition (CFO) and five degrees varus (medial wedge) with a 4 mm medial heel skive custom FOs condition (CVFO). A curve analysis, using 1D statistical parametric mapping (SMP), was used to assess differences in lower limb joint motion, joint moments and muscle activity over the stance phase of gait across conditions.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms located to the medial ankle or foot Pain on palpation to the posterior tibialis muscle tendon Positive single or double heel-rise test Foot flattening and ''too many toes" sign

Exclusion Criteria:

* Rigidity of those deformities Pain on palpation of the peroneal muscles Wearing any type of foot and/or ankle orthoses one month prior to the study onset History of corticosteroid injection in the tendon one month prior to the study onset Having a neurological disease or past history of surgery to the affected ankle

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Lower limbs' joint motion, joint moments and muscle activity | During the lab session
  A comparison of the lower limbs' joint motion, joint moments and muscle activity over the stance phase of gait between conditions
Comfort of the orthoses | During the lab session
  A comparison of the mean perceived comfort in each experimental condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Pavillon de l'Éducation Physique et des Sports - Université Laval, Québec, Canada

REFERENCES:
- [Background] Abousayed MM, Tartaglione JP, Rosenbaum AJ, Dipreta JA. Classifications in Brief: Johnson and Strom Classification of Adult-acquired Flatfoot Deformity. Clin Orthop Relat Res. 2016 Feb;474(2):588-93. doi: 10.1007/s11999-015-4581-6. No abstract available. PMID 26472584
- [Background] Barn R, Brandon M, Rafferty D, Sturrock RD, Steultjens M, Turner DE, Woodburn J. Kinematic, kinetic and electromyographic response to customized foot orthoses in patients with tibialis posterior tenosynovitis, pes plano valgus and rheumatoid arthritis. Rheumatology (Oxford). 2014 Jan;53(1):123-30. doi: 10.1093/rheumatology/ket337. Epub 2013 Oct 3. PMID 24097135
- [Background] Kulig K, Reischl SF, Pomrantz AB, Burnfield JM, Mais-Requejo S, Thordarson DB, Smith RW. Nonsurgical management of posterior tibial tendon dysfunction with orthoses and resistive exercise: a randomized controlled trial. Phys Ther. 2009 Jan;89(1):26-37. doi: 10.2522/ptj.20070242. Epub 2008 Nov 20. PMID 19022863
- [Background] Pataky TC. One-dimensional statistical parametric mapping in Python. Comput Methods Biomech Biomed Engin. 2012;15(3):295-301. doi: 10.1080/10255842.2010.527837. Epub 2011 Jul 14. PMID 21756121
- [Result] Chicoine D, Bouchard M, Laurendeau S, Moisan G, Belzile EL, Corbeil P. Biomechanical effects of three types of foot orthoses in individuals with posterior tibial tendon dysfunction. Gait Posture. 2021 Jan;83:237-244. doi: 10.1016/j.gaitpost.2020.11.001. Epub 2020 Nov 6. PMID 33190045